CLINICAL TRIAL: NCT04767945
Title: Registry of Adult Consenting Patients Admitted to the Liver Unit With Liver Cirrhosis
Brief Title: Cirrhosis Registry of Hospitalized Patients
Acronym: RH7
Status: Recruiting | Type: Observational
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Ľubomír Skladaný MD, PhD, Head, Department of Internal Medicine and HEGITO Liver Unit, Principal Investigator, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Other Study IDs: HEGITO2014
Record Dates: First submitted 2021-01-21; First posted 2021-02-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis, Liver; Frailty; Ascites; Encephalopathy; Infection
Keywords: Cirrhosis; decompensation; frailty
MeSH Terms: conditions — Liver Cirrhosis; Frailty; Ascites; Brain Diseases; Infections; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples Without DNA — Data collection is at times enriched by stool samples collection for 16SRNA microbiome analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with liver cirrhosis admitted to hospital liver unit: Consenting adults admitted with liver cirrhosis; recorded/uploaded are demographic, clinical, laboratory and imaging data

SUMMARY:
Cirrhosis registry of consecutive adult consenting patients hospitalized with liver cirrhosis in the tertiary liver unit

DETAILED DESCRIPTION:
On admission to F.D.Roosevelt Teaching Hospital / HEGITO Liver Unit (Div Hepatology, Gastroenterology and Liver Transplant), all the adult patients with liver cirrhosis are offered to participate.

After providing informed consent, their demographic, clinical and laboratory / imaging data are uploaded by dedicated study person After discharge from the hospital, follow-up is recommended and uploaded to RH7 (if the follow-up visits take place at this institution [FDR]) Mortality data are uploaded from the national registry of dead on regular basis

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis (primarily on clinical grounds)
* decompensating event leading to hospital admission
* informed consent

Exclusion Criteria:

* declined consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are patients with liver cirrhosis and indication for hospital admission who are or are not candidates for liver transplant and have or do not have liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of decompensation of liver cirrhosis | "1 year"
  Registrations reflect cirrhosis prevalence; decompensation are acute, chronic, or acute-on-chronic
Mortality | "1 year"
  Record mortality in registered cirrhotics

SECONDARY OUTCOMES:
Mortality | 90-day
  Record mortality in registered cirrhotics
Mortality | 1 year
  Record mortality in registered cirrhotics
Frailty | On admission
  Measurement of the liver frailty index

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Skladany, MD PhD, Principal Investigator — F.D.Roosevelt Teaching Hospital, Banska Bystrica, Slovakia
Locations (1):
- F.D.Roosevelt Teaching Hospital, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Sharing by request primarily by investigators from other centres, editors of medical journals, authors of meta analyses, etc
Supporting Information: Study Protocol, ICF, CSR
Time Frame: On request, immediately, open ended
Access Criteria: GDPR compliance Medical Journal Editorial office approved person Auditing authority Approved scientist
URL: http://www.fnspfdr.sk

REFERENCES:
- [Derived] Koller T, Vrbova P, Kubanek N, Zilincanova D, Selcanova SA, Havaj DJ, Skladany L. Assessment of intestinal inflammation via fecal calprotectin for early prediction of adverse outcomes in advanced chronic liver disease. United European Gastroenterol J. 2025 Apr;13(3):305-316. doi: 10.1002/ueg2.12633. Epub 2024 Jul 19. PMID 39031494